CLINICAL TRIAL: NCT01084460
Title: Follow-up of the Natural Course of the Small EUS-suspected Gastric Gastointestinal Stromal Tumors
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Hsiu-Po Wang, Department of Internal Medicine, National Taiwan University Hospital
Other Study IDs: 200812083R
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-03

CONDITIONS: Tumor
Keywords: Gastrointestinal stromal tumor,endoscopic ultrasound,submucosal tumor
MeSH Terms: conditions — Neoplasms; Gastrointestinal Stromal Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- EUS-suspected gastric GISTs: In this retrospective study, 50 patients with EUS-suspected gastric GISTs, less than 3 cm were enrolled and had EUS follow-up at least two times over a period of more than 24 months.

SUMMARY:
Gastric gastrointestinal stromal tumors (GISTs) less than 2 cm are usually followed up conservatively. However, little is known about the natural course of small GISTs. The goal of this study was to evaluate the clinical course of the small EUS-suspected gastric GISTs and to determine the size predicting subsequent progression with increased malignant potential.

ELIGIBILITY:
Inclusion Criteria:

* (1) a small tumor size, less than 3 cm;
* (2) patients declined surgical intervention at initial identification of the lesion;
* (3) at least two EUS follow-up procedures were recorded;
* (4) the EUS follow-up period was more than 24 months.

Exclusion Criteria:

* (1) a tumor size, larger than 3 cm;
* (2) less two EUS follow-up procedures were recorded;
* (3) the EUS follow-up period was less 24 months.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective study. We reviewed 256 consecutive patients with the diagnosis of suspected gastric GISTs by EUS, from January 1997 to December 2008 at the National Taiwan University Hospital, Yuan's General Hospital and En Chu Kong Hospital.
Sampling Method: Probability Sample
Dates: Start 1997-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hsiu Po Wang, MD, Principal Investigator — Department of Internal Medicine, National Taiwan University Hospital